CLINICAL TRIAL: NCT03509701
Title: Association Between Reversible Cerebral Vasoconstriction Syndrome and Herpes Zoster Infection
Brief Title: Reversible Cerebral Vasoconstriction Syndrome and Varicella Zoster Virus
Acronym: RCVS&VZV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Hanyang University (Other); Eulji University Hospital (Other); Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Prof., Asan Medical Center
Other Study IDs: 2018-0385
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Reversible Cerebral Vasoconstriction Syndrome; Varicella-zoster Virus Infection
Keywords: Reversible cerebral vasoconstriction syndrome; Herpes zoster; Varicella-zoster virus infection
MeSH Terms: conditions — Varicella Zoster Virus Infection; Herpes Zoster

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subject (RCVS): Patients who meet the definition of RCVS. (1) acute and severe headache with or without focal deficits or seizures, (2) uniphasic course without new symptoms more than 1 month after clinical onset, (3) segmental vasoconstriction of cerebral arteries shown by computed tomography angiography (CTA), magnetic resonance angiography (MRA) or transfemoral cerebral angiography (TFCA),(4) normal or near normal cerebrospinal fluid analysis and (5) complete or substantial normalisation of arteries shown by follow-up angiography within 12 weeks.
  Interventions: Diagnostic Test: VZV-specific antibody response from blood
- Control: Patients with thunderclap headache and intracranial stenosis, but not diagnosed as RCVS.
  Interventions: Diagnostic Test: VZV-specific antibody response from blood

INTERVENTIONS:
Diagnostic Test: VZV-specific antibody response from blood — Check VZV-specific antibody response, VZV specific T-cell mediated immune response by IFN-γ ELISPOT assay from blood, and real-time PCR results from saliva
  Other Names: VZV-specific T cell response from blood, viral load from saliva

SUMMARY:
Among patients with thunderclap headache who were admitted to the four participating hospitals, who has diffuse segmental vasoconstriction on CT angiography or MR angiography will be eligible for the study. Participants who meet the definition of RCVS will be enrolled as the case-patients and others will be enrolled as control-patients. The RCVS group will be defined when two or more neurologists agree by the clinical features and angiographic findings. The result of tests for varicella zoster virus titer will not be opened to neurologists until the end of the study. For case and control patients, tests for varicella zoster virus infection are (1) Pre-existing virological markers (ex. VZV-IgG, IgM, and VZV PCR in CSF or Skin lesion if present) (2) VZV-specific cell mediated immune response (CMI) at the time of admission and one month later (3) VZV in blood measured by quantitative test of viral load with real-time PCR and digital PCR for latent viral load (4) Quantitative test of viral load with real-time PCR in saliva at time of admission and one month later. Reactivation or infection of VZV of patients with RCVS and controls will be compared.

DETAILED DESCRIPTION:
In the previous pilot study, reactivation of VZV was confirmed in 63.6% of the patients as having RCVS by cell mediated immune response (CMI) test and 18.2% by Saliva PCR. None of patients who were simply stressed showed reactivation of VZV. Considering about 20% had false negative results in angiographic findings of RCVS, we set the effect size as 0.63 in group of subjects and 0.12 in group of controls. Using alpha values of 0.05 and beta values of 0.2, we calculated the target number of the study. If the ratio of cases to controls is 1:2, 9 case-patients and 18 control-patients were needed and if the ratio is 1:3, 8 case-patients and 24 control-patients were needed. We expect to enroll 10 case-patients and 20 to 30 control-patients within two years, considering the drop rate of 10~20%.

Baseline clinical information regarding age, sex, smoking history and medical comorbidities including hypertension (treated, systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at discharge), diabetes (treated, fasting blood glucose ≥126 mg/d), hyperlipidemia (treated, total cholesterol level ≥200 mg/dl or low-density lipoprotein level ≥140 mg/dl) and coronary artery disease will be collected on admission. Laboratory tests, including complete blood count, blood chemistry, c-reactive protein and erythrocyte sediment rate wil be performed. Images of brain MRI, MR angiography, CT angiography or digital substraction angiography will be gathered if present.

Tests for VZV specific antibody responses and T-cell mediated immune response will be performed by VZV specific ELISA and IFN-γ ELISPOT, respectively. Result for T cell responses will be shown as spot number per 10^6 PBMCs. On the day of blood sample collection, plasma will be isolated and freezed (-80℃). Peripheral mononuclear cells will be separated from the remaining blood samples and keep freezed (-190℃). Melt the frozen peripheral mononuclear cells and inoculate them on a plate (T-Track human IFN-γ, Lophius) with anti-human IFN-γ antibody and inoculate VZV lysate (Microbix) 50 ug/mL on them. After incubating 24 hours, the staining will be performed and the spot will be read in a automated ELISPOT reader (ELR07 reader system, Autoimmune Diagnostika GmbH).

For statistical analysis, patients with thunderclap headache will divided into two groups according to the presence of RCVS. Among them, the rate of infection with varicella zoster virus will be compared and analyzed. Fisher's exact test, Mann-Whitney test, Pearson correlation will be performed. Also, logistic regression analysis will be used, and covariates will be adjusted if needed. Sensitivity and specificity of tests for reactivation of VZV and RCVS will be analyzed too.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thunderclap headache and suspicious of intracranial vascular lesion by computed tomographic angiography (CTA) or magnetic resonance angiography (MRA).

Exclusion Criteria:

* Patients with life threatening medical condition
* Pregnant or scheduled for pregnancy
* Unwilling or unable to give informed consent
* Patients who confirmed vasculitis
* Patients with genetic disease for vascular disorder

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited Asan medical center, Hanyang University Guri Hospital, Nowon Eulji Medical Center, or Kangbuk Samsung Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Infection or reactivation of varicella zoster virus (VZV) | At the time of enrolled.
  Compare prevalence of infection or reactivation of VZV in case-patients and control-patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD.Phd, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singhal AB, Hajj-Ali RA, Topcuoglu MA, Fok J, Bena J, Yang D, Calabrese LH. Reversible cerebral vasoconstriction syndromes: analysis of 139 cases. Arch Neurol. 2011 Aug;68(8):1005-12. doi: 10.1001/archneurol.2011.68. Epub 2011 Apr 11. PMID 21482916
- [Background] Katz BS, Fugate JE, Ameriso SF, Pujol-Lereis VA, Mandrekar J, Flemming KD, Kallmes DF, Rabinstein AA. Clinical worsening in reversible cerebral vasoconstriction syndrome. JAMA Neurol. 2014 Jan;71(1):68-73. doi: 10.1001/jamaneurol.2013.4639. PMID 24190097
- [Background] Miller TR, Shivashankar R, Mossa-Basha M, Gandhi D. Reversible Cerebral Vasoconstriction Syndrome, Part 1: Epidemiology, Pathogenesis, and Clinical Course. AJNR Am J Neuroradiol. 2015 Aug;36(8):1392-9. doi: 10.3174/ajnr.A4214. Epub 2015 Jan 15. PMID 25593203
- [Background] Cuvinciuc V, Viguier A, Calviere L, Raposo N, Larrue V, Cognard C, Bonneville F. Isolated acute nontraumatic cortical subarachnoid hemorrhage. AJNR Am J Neuroradiol. 2010 Sep;31(8):1355-62. doi: 10.3174/ajnr.A1986. Epub 2010 Jan 21. PMID 20093311
- [Background] Kwon SU, Yun SC, Kim MC, Kim BJ, Lee SH, Lee SO, Choi SH, Kim YS, Woo JH, Kim SH. Risk of stroke and transient ischaemic attack after herpes zoster. Clin Microbiol Infect. 2016 Jun;22(6):542-8. doi: 10.1016/j.cmi.2016.03.003. Epub 2016 Mar 16. PMID 26992774
- [Background] Kim MC, Yun SC, Lee HB, Lee PH, Lee SW, Choi SH, Kim YS, Woo JH, Kim SH, Kwon SU. Herpes Zoster Increases the Risk of Stroke and Myocardial Infarction. J Am Coll Cardiol. 2017 Jul 11;70(2):295-296. doi: 10.1016/j.jacc.2017.05.015. No abstract available. PMID 28683973
- [Background] Bartynski WS, Boardman JF, Zeigler ZR, Shadduck RK, Lister J. Posterior reversible encephalopathy syndrome in infection, sepsis, and shock. AJNR Am J Neuroradiol. 2006 Nov-Dec;27(10):2179-90. PMID 17110690
- [Background] Park SY, Kim JY, Kim JA, Kwon JS, Kim SM, Jeon NY, Kim MC, Chong YP, Lee SO, Choi SH, Kim YS, Woo JH, Kim SH. Diagnostic Usefulness of Varicella-Zoster Virus Real-Time Polymerase Chain Reaction Analysis of DNA in Saliva and Plasma Specimens From Patients With Herpes Zoster. J Infect Dis. 2017 Dec 27;217(1):51-57. doi: 10.1093/infdis/jix508. PMID 29029120
- [Background] Yancy H, Lee-Iannotti JK, Schwedt TJ, Dodick DW. Reversible cerebral vasoconstriction syndrome. Headache. 2013 Mar;53(3):570-6. doi: 10.1111/head.12040. PMID 23489219
- [Background] Ducros A. Reversible cerebral vasoconstriction syndrome. Lancet Neurol. 2012 Oct;11(10):906-17. doi: 10.1016/S1474-4422(12)70135-7. PMID 22995694